CLINICAL TRIAL: NCT00197366
Title: Development of Resistance Mutations in the Human Immunodeficiency Virus (HIV) in Pregnant HIV+ Women Receiving Perinatal Antiretroviral Therapy in Israel
Brief Title: Development of Resistance Mutations in Pregnant HIV-positive (+) Women Following Perinatal Antiretroviral Therapy in Israel
Status: Terminated | Type: Observational
Why Stopped: Difficulties in data collection
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 16-25.02.05-HMO-CTIL
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: pregnancy; HIV-positive; HIV resistance; HIV
MeSH Terms: conditions — HIV Infections; HIV Seropositivity

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
It has been shown that treatment of HIV-positive women with antiretroviral medication during pregnancy reduces the risk of HIV transmission to the child. However, such treatment could lead to the selection of resistant virus strains in the mother. The object of this study is to check HIV+ pregnant women for resistance mutations in HIV before and after the antiretroviral therapy they receive during pregnancy. HIV-positive newborns will also be tested, to see if a resistant virus strain was transmitted from mother to child.

DETAILED DESCRIPTION:
The project will be performed in collaboration with the Israeli National HIV Reference Center Laboratory, which maintains a national bank of HIV-positive blood samples, and with HIV/AIDS treatment centers located throughout Israel.

An initial survey will identify retrospectively those HIV+ women who were given antiretroviral therapy while pregnant and stopped treatment after delivery. The list of HIV+ deliveries over the past five years in each participating hospital will be reviewed, and all HIV-positive women who received antiretroviral treatment during pregnancy will be invited to participate in the study project. Women who are currently pregnant, or become pregnant during the study, will be invited to participate when pregnancy is diagnosed. After obtaining informed consent, two blood samples will be obtained: one before the initiation of perinatal treatment, and the other following delivery. (Due to technical limitations, only samples with viral loads above 1000 cp/ml can be genotyped. It is expected that HIV loads will rise following cessation of antiretroviral treatment, and that almost all samples will be eligible for resistance testing.)

In addition, after obtaining maternal informed consent, samples from newborns infected perinatally with HIV will also be tested for resistance mutations, and these will be compared with the resistance pattern found in the mother.

The samples obtained will be tested for genotypic resistance mutations. The results will be transmitted to the treating physician to assist in choice of antiretroviral therapy for the women and their children, if needed. The data will also be used to establish a national database to evaluate and improve existing protocols for perinatal antiretroviral treatment, and will be used to contribute to international databases of HIV resistance. All resistance data, except that given to the health care provider(s), will be transmitted without additional identifying information.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-positive women currently pregnant or with a past pregnancy in Israel
2. Blood/plasma samples available before and/or after perinatal antiretroviral treatment (before or during pregnancy if not treated)
3. HIV viral load in the samples adequate for resistance testing (approximately 1000 copies/ml)
4. Informed consent obtained

Exclusion Criteria:

1. Samples not available or inadequate viral load
2. Informed consent not obtained

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-03; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Maayan, MD, Principal Investigator — Hadassah-Hebrew U Medical Center; Zehava Grossman, PhD, Principal Investigator — Central Virology Laboratory Tel HaShomer; Rebekah Karplus, MD, Principal Investigator — Hadassah-Hebrew U Medical Center
Locations (5):
- Israel (5):
  - Soroka University Medical Center, Beersheva
  - Rambam Medical Center, Haifa
  - AIDS Center, Hadassah-Hebrew U Medical Organisation, Jerusalem
  - Meir Hospital Sapir Medical Center, Kfar Saba
  - Kaplan Medical Center, Rehovot